CLINICAL TRIAL: NCT02109302
Title: Identification Des Bases moléculaires de l'éjaculation prématurée Primaire
Brief Title: Primary Premature Ejaculation Genetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C12-32; 2012-A01055-38 (Registry Identifier: ID RCB)
Record Dates: First submitted 2014-04-02; First posted 2014-04-09 (Estimated); Last update posted 2025-03-14 (Actual); Status verified 2025-01

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Men over 18 years of age with primary Premature Ejaculation (Experimental)
  Interventions: Procedure: Blood sample; Procedure: Skin biopsy; Other: Questionnaire

INTERVENTIONS:
Procedure: Blood sample
Procedure: Skin biopsy
Other: Questionnaire

SUMMARY:
The main objective of our study is to identify the first genetic etiology of primary Premature Ejaculation (PE). We will test and evaluate the existence of genetic determinism conferring susceptibility to a life-long syndrome (primary premature ejaculation) in some patients. To this end, we plan to establish a collection of biological samples and a database of patients with this extreme syndrome, which we will analyze by Genome Wide analysis. This will lead to improvements in the biological understanding, the "knowledge" of physicians of the disease, and should improve the patients' quality of life. Not all PE cases have the same physiopathology and treatment efficiency, which depend on the specific mechanism involved in the clinical context. Our work will make it possible to develop new therapeutic approaches suitable for a large proportion of individuals presenting PE. This integrative approach combining researchers, patients and ethics committees will facilitate profound reflection, promoting the creation of suitable structures capable of receiving patients for appropriate consultations. This unique study of PE should also favor industrial partnerships.

DETAILED DESCRIPTION:
2.1 Main Objective

* To identify the molecular basis of primary premature ejaculation (PPE) in humans for the development of new adapted therapy.
* Check and confirm the genetic hypothesis of PPE to fill the void of genetic knowledge about this syndrome.
* Improve knowledge of physicians on this disease to increase the comfort of life of patients.

2.2 Secondary Objectives

* Provide the basis for new therapeutic approaches.
* Expanded knowledge of the aetiology of PE and allow better management of patients.
* Develop strategies to prevent the consequences, sometimes severe , of this condition on the intimate, personal, social and professional life of these patients. Because all the PE do not have the same pathophysiology and treatment success depends on its relevance to the specific mechanism of the clinical form concerned.
* Increase the comfort of life of the patients.
* Eliminate public prejudice based on misconceptions.

ELIGIBILITY:
Inclusion Criteria:

1. . Patients (index cases ) Prospective and retrospective cases

   * Man aged over 18 years
   * signing the informed consent
   * Presenting primary PE
   * have an affiliation to a social security system
2. . Related

   * Male or female over 18 years
   * be related to the index case
   * signing the informed consent
   * have an affiliation to a social security system

Non Inclusion Criteria:

1. . Patients ( index case ) :

   * Be aged under 18
   * have known genetic variations that predispose or can promote psychological disorders that can lead to PE ( eg: Kallman 's Syndrome , micropenis , testicular dysgenesis , Klinfelter syndrome, Leydig cell hypoplasia )
   * have had psycho- social and psycho- traumatic factors in childhood
   * Inability to receive clear information on the protocol
   * Person deprived of liberty by judicial or administrative decision
   * Major Person subject of legal protection or unable to consent
   * Refusal to be informed of an abnormality detected after genetic testing
   * History of allergies to lidocaine or other anesthetic agent used during puncture or blood sample
2. . Related :

   * Age <18 years
   * Inability to receive clear information about the protocol . Unable to participate in the entire study.
   * No coverage by the social security system
   * Absence of signature of consent or refusal of the related party
   * Person deprived of liberty by judicial or administrative decision
   * Major Person subject of legal protection or unable to consent
   * Refusal to be informed of a genetic abnormality detected
   * History of allergies to lidocaine or other anesthetic agent used during puncture or blood sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with genetic mutations of susceptibility to primary PE | 4 years
  We will perform WES (Whole Exome Sequencing) to identify shared defective genes in 20 patients. In case of genetic uniformity and of a genetically homogeneous recruitment, we hope to highlight such a gene in several individuals. As primary PE are very rare, this group should have defective genes at much higher frequencies than in the control population (NCBI, 1000 genome and housing-genome). This will allow us to identify genetic mutations of susceptibility to primary PE.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Alcaïs, MD, Principal Investigator — Hôpital Necker
Locations (3):
- France (3):
  - Polyclinique de Blois, La Chaussée-Saint-Victor
  - Hôpital Saint Joseph, Marseille
  - Hôpital Necker, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Porto R, Giuliano F. [Premature ejaculation]. Prog Urol. 2013 Jul;23(9):647-56. doi: 10.1016/j.purol.2013.01.005. Epub 2013 Mar 1. French. PMID 23830259